CLINICAL TRIAL: NCT01560741
Title: Randomized Trial Comparing Telemedicine Monitoring and Titration in Patients Initiating Non-invasive Ventilation With Usual Care (TELEMOTINIV Study)
Brief Title: Telemedicine and Ventilator Titration in Chronic Respiratory Patients Initiating Non-invasive Ventilation
Acronym: TeleMotiNIV
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, Miguel R. Goncalves, Clinical Professor, Hospital Sao Joao
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TeleMotiNIV2012
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Neuromuscular Disease; Chest Wall Disorders; Obesity Hypoventilation Syndrome
Keywords: Chronic respiratory failure; Noninvasive Mechanical Ventilation; Home-care; Telemedicine; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neuromuscular Diseases; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine Group (Active Comparator): Patients will be initiated and adapted on non-invasive home mechanical ventilation in Pulmonology Department of S. João Hospital, in an outpatient setting, according to the prevailing standard of care for Chronic Respiratory Diseases patients in this unit. Patients will be provided with a ventilator outfitted with a wireless transmitter to allow the remote data collection of compliance and efficacy information. While patient sleeps, data is collected. If abnormalities criteria will be detected, remote titration of ventilator settings will be done to optimise therapy. Patient will be monitored again and data analyzed. This procedure will be repeated until we obtained the optimal ventilator parameters for each patient in this group. Nocturnal oximetry under home mechanical non-invasive ventilation will be carried out after one week and one month of treatment. Subjects also receive pre-arranged telephone calls to assist with progress.
  Interventions: Device: Telemonitoring tools
- Usual care (Other): Patients will be initiated and adapted on non-invasive home mechanical ventilation in Pulmonology Department of S. João Hospital, in an outpatient setting, according to the prevailing standard of care for Chronic Respiratory Diseases patients in this unit. Patients will be assessed by a hospital visit scheduled at the end of third month after their initial adaptation. In this hospital visit data provided by the ventilator will be transferred to research team computer so they could evaluate patient compliance and efficacy of ventilation criteria under the parameters used at home present at the time of assessment. If abnormality criteria will be detected, re-titration of ventilator settings will be made. Patients will be encouraged to call their respiratory consultant any time they had a problem or concern.
  Interventions: Device: Usual Care

INTERVENTIONS:
Device: Telemonitoring tools — Patients will go home with telemedicine tools to monitor efficacy and compliance of non-invasive home mechanical ventilation
  Other Names: wireless transmiter
  Arms: Telemedicine Group
Device: Usual Care — The assessment of efficacy and compliance will be monitor at the end of third month. This is the date of the scheduled hospital visit.
  Other Names: Hospital visit
  Arms: Usual care

SUMMARY:
The critical nature of respiratory diseases, the continuously increasing prevalence of these conditions, and the subjective perception of patients vis-à-vis their pulmonary function and health status underscore the importance of home telemonitoring. These conditions are critical and necessitate close and regular monitoring that may be achieved at distance using telemonitoring. This study will assess a number of measures both at baseline and post-intervention from a number of domains, including Arterial Blood Gases (ABG), BiPAP-related data, chronic respiratory failure symptoms, health-related quality of life, patients satisfaction and utilization of healthcare resources.

DETAILED DESCRIPTION:
In recent years home care is becoming increasingly used and considered by some the future of healthcare. Home mechanical ventilation has been shown to improve morbidity and mortality in patients with chronic respiratory failure of different aetiologies. A French survey suggests an increase of 12% of cases per year. With the prospect of a substantial increase of ventilated patients at home, facilities and resources have not been proportionally growing, so new approaches should be investigated and addressed to absorb this constant flux of patients.

Telemedicine is defined as the broad use of electronic and communications technologies to provide and support remote monitoring of health status. It has been shown to be an effective alternative model of care for managing chronic diseases. It as also been shown to reduce healthcare costs and is a major topic on the agendas of health and social care policies in Europe.

Home telemonitoring of respiratory conditions results in early identification of deteriorations in patient condition and symptom control.

However, evidence on the magnitude of clinical and structural effects remains preliminary, with variations in study approaches and an absence of robust study designs and formal evaluations.

The objective is gathering data that can be help to establish guidelines for non invasive home mechanical ventilation initiation and quality control.

ELIGIBILITY:
Inclusion Criteria:

OHS:

* PaCO2 > 45 mmHg;
* IMC > 40 Kg/m2

COPD:

* Age < 80 years;
* Receiving appropriate medical therapy according to gold guidelines
* Long-term oxygen therapy (LTOT) for at least 3 months;
* PaCO2 > 50 mmHg during room air
* ph > 7,35 and free from exacerbations in the 4 weeks preceding recruitment;
* One exacerbation in the last year before preceding recruitment with necessity of NIV in the acute care setting;
* FEV1 < 1,5l or < 50% predicted;
* FEV1/FVC < 60%
* Total Lung Capacity (TLC)≥ 90% predicted;
* PaO2 < 60 mmHg breathing room air at rest.

NMD and CWD:

* PaCO2 > 45 mmHg;
* Significant nocturnal desaturation
* FVC < 50% predicted;
* SNIP < 40 cmH20
* MIP < 60% predicted
* Ortopnea;
* 20% drop of VC in supine position.

Exclusion Criteria:

OHS:

* COPD
* NMD

COPD:

* 15% increase in FEV1 after inhaled Salbutamol (200 µg);
* Active smoking;
* History of OSA (with AHI > 15 episodes.h-1)

NMD and CWD:

* COPD;
* OHS;
* PCF < 270;
* Severe bulbar weakness (ALSFRS bulbar subscore 0-3)
* MIC/VC=1

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Nocturnal noninvasive ventilation compliance per day | 9 months
  We aim to detect a difference of 1 hour in the mean of nightly hours of use, assuming a standard deviation (SD) of 2 hours.

SECONDARY OUTCOMES:
Health Economics Evaluation | 9 months
  This project project will randomize 2 distinct groups adopting different tecnhologies so we will be able to quantify the economic/budget impacts for each alternative
Health related Quality of Life | 9 months
  Incremental gains in quality of life will be evalueted from a clinical perspective and as an investment.
Arterial Blood Gases | 9 months
  We aim to detect a

CONTACTS AND LOCATIONS:
Overall Officials: J C Winck, Phd, Principal Investigator — Hospital de S. João
Locations (1):
- Hospital de S.João, Porto, Porto District, Portugal